CLINICAL TRIAL: NCT05840315
Title: Feasibility of High Density Sit-to-stand Functional Resistance Training in Patients with Hip Fracture. a Non-randomized Pilot Trial
Brief Title: Feasibility of High Density Sit-to-stand Functional Resistance Training in Patients with Hip Fracture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Horsholm Municipality (Other)
Responsible Party: Principal Investigator, Niklas Grundt Hansen, Research Therapist, Horsholm Municipality
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RSS protokol Hoftefrak
Record Dates: First submitted 2023-03-22; First posted 2023-05-03 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Hip Fractures; Sarcopenia; Fall Injury
Keywords: physical therapy; resistance training
MeSH Terms: conditions — Hip Fractures; Sarcopenia | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Three stages of single arm non-randomized feasibility trial set-up, testing an interventions feasibility, combined with the usual rehabilitation program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 1 (Experimental): First subtrial (participants 1-10):
  Sit-to-stand-to-sit training
  Interventions: Dietary Supplement: Basic intervention and nutritional intervention; Procedure: Sit-to-stand
- Phase 2 (Experimental): Second subtrial (participants 11-20):
  Sit-to-stand and leg press training.
  Interventions: Dietary Supplement: Basic intervention and nutritional intervention; Procedure: Sit-to-stand; Procedure: Leg press
- Phase 3 (Experimental): Third subtrial (participants 21-30):
  Sit-to-stand and hip abduction training.
  Interventions: Dietary Supplement: Basic intervention and nutritional intervention; Procedure: Sit-to-stand; Procedure: Hip abduction

INTERVENTIONS:
Dietary Supplement: Basic intervention and nutritional intervention — The training plan is divided into 3 parts with different sub-components. There will be ongoing enrollment until 10 participants have been recruited, after which the next sub-trial will start recruitment. The intervention from the respective sub-trials is described in the individual study phases.
  Participants attend one-hour exercise sessions, 2 times/week for 8 weeks, in groups of 4-7 patients, supervised by 2-3 physio therapists.
  After completion of the physical intervention all participants are given a nutritional supplement, being a 200ml cocoa(Chokolate milk), containing 7 grams of protein, 24grams of carbohydrates, 5 grams of fat and in total 166 kilocalories. If any participant has lactose intolerance or diabetes, they are advised to bring an egg and a piece of rye bread to secure an equal amount of protein and calories.
  Other Names: Nutritional intervention
Procedure: Sit-to-stand — First subtrial (participants 1-10):
  Sit-to-stand-to-sit training: Participants will be instructed to do as many sit-to-stand repetitions as possible without using their arms in a 30 second window, followed by a 30 second rest. This sequence is repeated for a total of 10 sets (a total of 10 minutes). Standard seat height of chair is 46 cm.
  Progression/regression: If a participant is unable to do at least 6 repetitions on the first sit-to-stand test, they are allowed to sit on a 6cm airex pillow while performing the exercise. When a single set of 12 chair rises are attained or total amount of repetitions reach 100 in 10 sets on an airex, the participant progresses to sitting on a 6-0,5cm wedge pillow, and again when the participant attains 12 rises, he/she progress to rising from the standard chair height.
  Other Names: Resistance training
Procedure: Leg press — Second subtrial (participants 11-20):
  In addition to the above intervention, progressive strength training is performed on a leg press, consisting of 3 sets of 8-12RM. Participants are instructed to do as many repetitions as possible, and the weight is increased if either 12 repetitions are performed on three consecutive sets or a single set or more than 14 repetitions are completed. If fewer than 6 repetitions are performed, the weight is reduced . There is a minimum of one minute break between each set of training on the leg press.
  Other Names: Resistance training
  Arms: Phase 2
Procedure: Hip abduction — Third subtrial (participants 21-30):
  In addition to interventions described in sub-trial 1, Third subtrial will perform progressive strength training for the gluteal muscles is carried out in form of hip abduction, using rubber bands, consisting of 3 sets of 8-12RM using the same procedure as above mentioned for the leg press.
  Hip abduction will be performed from a standing position with a straight arm length from a wall, supporting the wall. The participant will be instructed to abduct the hip facing the wall until the foot is in contact with the wall, and then back until it touches the standing leg.
  Progression will be placing a rubber band just proximal to the knee with resistances being: yellow= light, red= moderate, blue= heavy.
  further progression will be placing the rubber band around the ankles using the same progression as above.
  Other Names: Resistance training
  Arms: Phase 3

SUMMARY:
The objective of this study is to examine if functional high-density, high-volume chair rise training is feasible for increasing lower extremity strength without causing excessive hip pain during execution in patients with hip fracture following a municipality -based outpatient rehabilitation program.

Feasibility criteria is defined as: 1) hip fracture-related pain might increase during the exercise programme, but not persistent after each session. 2) adherence to the program must be 75% or more. 3) Less than 20% drop-outs due to pain and/or discomfort during training.

DETAILED DESCRIPTION:
Background and rationale:

Hip fractures are associated with decrease in muscle strength, Rehabilitation after hip fractures typically include types of resistance training, functional training and cardiovascular training Factors affecting the functional prognosis after hip fracture surgery are multiple, and patients are at risk of decreased physical function new injurious falls and fractures and increased need of supportive care.

Earlier research has shown that daily on weekdays, progressive knee-extension strength training (three sets with a 10RM load) is a feasible and potentially effective treatment for increasing muscle strength in patients with hip fractures when commenced few days after surgery.

Extended physical therapy including strength training implemented about 6 weeks or later after hip fracture surgery seem to promote recovery of physical function.

The goal of rehabilitation is to reach the highest degree of autonomy as possible, which in sarcopenic older adults requires increasing the muscle strength in the lower extremities. Higher volume resistance training has been associated with increased muscle mass and strength in both young and older populations Resistance training for elderly patients is usually done to failure to ensure adequate volume for muscle hypertrophy and strength increases.

In comparison, Sit-to-stand chair exercises has earlier been executed as progressive training and shows promising results as to increasing ability to rise from a lower chair In stroke patients. Sit-to-stand exercise has been shown to be a good whole body exercise and with effects of the exercises ranging from increased leg strength to association with lower degree of dysphagia in stroke patients, when done in addition to the convalescence rehabilitation program.

To the researchers knowledge there exist no other trials testing systematic use of very high training volume of sit-to-stand exercises in rehabilitation of older patients with hip fractures.

This trial searches to combine training with high volume of sit-to-stand exercises with training to volitional failure on leg press and hip abductions to employ combinations of heavy, progressive resistance training and very high volume of total training (29 sets per week) Objectives The objective of this study is to examine if functional high-density, high-volume chair rise training is feasible for increasing lower extremity strength without causing excessive hip pain during execution in patients with hip fracture following a municipality -based outpatient rehabilitation program.

Feasibility criteria is defined as: 1) hip fracture-related pain might increase during the exercise programme, but not persistent after each session. 2) adherence to the program must be 75% or more. 3) Less than 20% drop-outs due to pain and/or discomfort during training.

ELIGIBILITY:
Study setting Training and data collection will be executed at a rehabilitation centre in Hørsholm municipality, capital region, Denmark.

Eligibility criteria Patients with hip fractures having

* Referred to rehabilitation due to hip fracture
* Age of 60 years or older
* Cumulated Ambulation Score 5 or higher

Exclusion criteria

* Moderate to severe dementia
* Patients suffering from a severe medical condition not allowing them to follow a physical exercise program
* Cancer
* Alcohol intake >21/14 units a week for men/women.
* Patients not allowed full weight bearing on the fractured leg
* Patients with 2 Hansson pins or similar procedure for cervical femoral fractures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the interventions; Adherence | Measured during the 8 week intervention
  Feasibility is evaluated based on adherence to the program. Adherence to the program must be 75% or more, and drop outs due to pain or discomfort during training should be no more than 20%.
Tolerability of the interventions; Hip fracture related pain | Measured during the 8 week intervention
  Hip fracture-related pain during exercise, and dropouts. Hip fracture-related pain should not increase to more than a maximum of 3 VRS points (severe pain) during exercise and reduced thereafter, Patient rating pain on a verbal rating scale of 0-4 0: no pain, 1: slight pain, 2: Moderate pain, 3: severe pain and 4: Unbearable pain.

SECONDARY OUTCOMES:
Sit-to-stand- test | Baseline(within the first week before starting the intervention) and immediately post intervention period
  Change in the number of times the patient comes to full standing position in 30 seconds from a chair with a seat height of 44-47cm. The Sit to Stand test provides a measurement of a person's lower body (particularly quadriceps) strength(18). Hip-pain will be assessed before and after (describing the maximum pain during testing) testing with the VRS (17).
Change in 10m walk test, using regular walk speed and standing start. | Baseline(within the first week before starting the intervention) and immediately post intervention period
  The time it takes the patient to walk 10 meters with a standing start, using walking aid if needed (19). The 10m. walk test gives an indication of a person's ability to walk and is recommended in the sarcopenia screening algorithm (20).
Change in Handgrip strength | Baseline(within the first week before starting the intervention) and immediately post intervention period
  The maximum grip force a person can apply to a handheld dynamometer, defined as the highest of three maximum efforts (up to five) with the dominant hand. Handgrip strength is associated with total upper body strength and is recommended in the sarcopenia screening algorithm(18,20)
SARC-F questionnaire | Baseline(within the first week before starting the intervention) and immediately post intervention period
  The Sarc-F is a 5-item questionnaire subjectively assessing strength, ability to walk, rise from a chair, walking on stairs and how often a person falls. Sarc-F is associated with the prevalence of sarcopenia and is the first test in the sarcopenia screening algorithm (20).
Prevalence and severity of sarcopenia | Baseline(within the first week before starting the intervention) and immediately post intervention period
  Sarcopenia is defined according to the European guidelines EWSGOP2 (20), based on low muscle strength (measured as Handgrip strength or STS test), Low muscle mass (measured with bioimpedance) and low muscle function (measured with 10m walk test or other performance tests )(20).
New mobility score | Baseline(within the first week before starting the intervention) and immediately post intervention period,(including pre-fracture by recall)
  New Mobility Score assesses walking function; indoor, outdoors and during shopping. 0-3 points are given for each function, resulting in a score ranging from 0-9 points. A change of 1 point is considered as clinically relevant change. New mobility score is a strong predictor of mortality and other outcomes after hip fracture (21,22).
Falls Efficacy Scale-International | Baseline(within the first week before starting the intervention) and immediately post intervention period
  Falls Efficacy Scale-International is a measure of "concerns about falling" intended to be used in an adult and elderly population. It is a 16 item questionnaire, useful to the researchers and clinicians interested in fear of falling, with a score ranging from minimum 16 (no concern about falling) to maximum 64 (severe concern about falling) (23).
Quality of life by EQ5D-5L | Baseline(within the first week before starting the intervention) and immediately post intervention period
  Assessment of quality of life using the EQ-5D-5L. EQ-5D is a non-disease-specific (generic) instrument developed to assess health-related quality of life. Rating instrument based on self-assessment of one's own condition. The EQ-5D is a widely used generic health-related quality of life instrument that has been used to describe population health and health outcomes in clinical trials and health economic evaluations
Quality of life by EQ-VAS | Baseline(within the first week before starting the intervention) and immediately post intervention period
  Assessment of quality of life using the EQ-VAS. EQ-5D is a non-disease-specific (generic) instrument developed to assess health-related quality of life. Rating instrument based on self-assessment of one's own condition. The EQ-5D is a widely used generic health-related quality of life instrument that has been used to describe population health and health outcomes in clinical trials and health economic evaluations

OTHER OUTCOMES:
BMI (kg/m2) | Baseline(within the first week before starting the intervention) and immediately post intervention period
  body weight in kg will be measured on a regular scale and to the nearest 100 grams. Participants will be weighed without shoes and with as little clothes as possible. Height will be measured on bare feet with a yardstick fixed to the wall and to the nearest cm. There will be determined if lower BMI or muscle mass results in less effect of an physical therapy intervention.
Body composition | Baseline(within the first week before starting the intervention) and immediately post intervention period
  Changes in body composition (muscle mass) during the intervention. Body composition will be determined on at Tanita scale, measuring body composition via bioimpedance. There will be determined if lower BMI or muscle mass results in less effect of an physical therapy intervention.
Home care | Measured pre-fracure (by recall), Baseline, immediately post intervention period and after 3 and 6 months after completing the intervention.
  The amount of hours dedicated to home care on a weekly basis from pre-fracture, at enrollment of intervention and after the end of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Grundt Hansen, Msc. PT, Principal Investigator — Research therapist, Hørsholm municipality, capital region; Morten Ta Kristensen, Professor, Study Director — Department of Physical and Occupational Therapy, Bispebjerg and Frederiksberg hospitals, Denmark
Locations (1):
- Hørsholm municipality, Hørsholm, Capitol Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kronborg L, Bandholm T, Palm H, Kehlet H, Kristensen MT. Feasibility of progressive strength training implemented in the acute ward after hip fracture surgery. PLoS One. 2014 Apr 3;9(4):e93332. doi: 10.1371/journal.pone.0093332. eCollection 2014. PMID 24699276
- [Background] Kristensen MT, Bandholm T, Bencke J, Ekdahl C, Kehlet H. Knee-extension strength, postural control and function are related to fracture type and thigh edema in patients with hip fracture. Clin Biomech (Bristol). 2009 Feb;24(2):218-24. doi: 10.1016/j.clinbiomech.2008.10.003. Epub 2008 Dec 16. PMID 19091449
- [Background] Overgaard J, Kristensen MT. Feasibility of progressive strength training shortly after hip fracture surgery. World J Orthop. 2013 Oct 18;4(4):248-58. doi: 10.5312/wjo.v4.i4.248. eCollection 2013. PMID 24147260
- [Background] Hulsbaek S, Juhl C, Ropke A, Bandholm T, Kristensen MT. Exercise Therapy Is Effective at Improving Short- and Long-Term Mobility, Activities of Daily Living, and Balance in Older Patients Following Hip Fracture: A Systematic Review and Meta-Analysis. J Gerontol A Biol Sci Med Sci. 2022 Apr 1;77(4):861-871. doi: 10.1093/gerona/glab236. PMID 34387664
- [Background] Kristensen MT. Factors affecting functional prognosis of patients with hip fracture. Eur J Phys Rehabil Med. 2011 Jun;47(2):257-64. PMID 21597435
- [Background] Rosell PA, Parker MJ. Functional outcome after hip fracture. A 1-year prospective outcome study of 275 patients. Injury. 2003 Jul;34(7):529-32. doi: 10.1016/s0020-1383(02)00414-x. PMID 12832181
- [Background] Ariza-Vega P, Jimenez-Moleon JJ, Kristensen MT. Change of residence and functional status within three months and one year following hip fracture surgery. Disabil Rehabil. 2014;36(8):685-90. doi: 10.3109/09638288.2013.813081. Epub 2013 Aug 6. PMID 23919643
- [Background] Egan M, Jaglal S, Byrne K, Wells J, Stolee P. Factors associated with a second hip fracture: a systematic review. Clin Rehabil. 2008 Mar;22(3):272-82. doi: 10.1177/0269215507081573. Epub 2007 Dec 5. PMID 18057086
- [Background] Auais MA, Eilayyan O, Mayo NE. Extended exercise rehabilitation after hip fracture improves patients' physical function: a systematic review and meta-analysis. Phys Ther. 2012 Nov;92(11):1437-51. doi: 10.2522/ptj.20110274. Epub 2012 Jul 19. PMID 22822235
- [Background] Fragala MS, Cadore EL, Dorgo S, Izquierdo M, Kraemer WJ, Peterson MD, Ryan ED. Resistance Training for Older Adults: Position Statement From the National Strength and Conditioning Association. J Strength Cond Res. 2019 Aug;33(8):2019-2052. doi: 10.1519/JSC.0000000000003230. PMID 31343601
- [Background] Schoenfeld BJ, Ogborn D, Krieger JW. Dose-response relationship between weekly resistance training volume and increases in muscle mass: A systematic review and meta-analysis. J Sports Sci. 2017 Jun;35(11):1073-1082. doi: 10.1080/02640414.2016.1210197. Epub 2016 Jul 19. PMID 27433992
- [Background] Borde R, Hortobagyi T, Granacher U. Dose-Response Relationships of Resistance Training in Healthy Old Adults: A Systematic Review and Meta-Analysis. Sports Med. 2015 Dec;45(12):1693-720. doi: 10.1007/s40279-015-0385-9. PMID 26420238
- [Background] Nobrega SR, Libardi CA. Is Resistance Training to Muscular Failure Necessary? Front Physiol. 2016 Jan 29;7:10. doi: 10.3389/fphys.2016.00010. eCollection 2016. No abstract available. PMID 26858654
- [Background] de Sousa DG, Harvey LA, Dorsch S, Varettas B, Jamieson S, Murphy A, Giaccari S. Two weeks of intensive sit-to-stand training in addition to usual care improves sit-to-stand ability in people who are unable to stand up independently after stroke: a randomised trial. J Physiother. 2019 Jul;65(3):152-158. doi: 10.1016/j.jphys.2019.05.007. Epub 2019 Jun 18. PMID 31227279
- [Background] Yoshimura Y, Wakabayashi H, Nagano F, Bise T, Shimazu S, Shiraishi A. Chair-stand exercise improves post-stroke dysphagia. Geriatr Gerontol Int. 2020 Oct;20(10):885-891. doi: 10.1111/ggi.13998. Epub 2020 Aug 9. PMID 32772455
- [Background] Kristensen MT, Foss NB. Danish version of Verbal Rating Scale (VRS 0-4 points) - Verbal Rang Skala (VRS). [Internet]. Unpublished; 2020 [henvist 7. marts 2023]. Tilgængelig hos: http://rgdoi.net/10.13140/RG.2.2.19739.41769/2
- [Background] Bech RD, Lauritsen J, Ovesen O, Overgaard S. The Verbal Rating Scale Is Reliable for Assessment of Postoperative Pain in Hip Fracture Patients. Pain Res Treat. 2015;2015:676212. doi: 10.1155/2015/676212. Epub 2015 May 20. PMID 26078880
- [Background] Kristensen MT, Dall CH, Aadahl M, Suetta C. Systematic assessment of physical function in adult patients across diagnoses. Ugeskr Laeger. 2022 Oct 24;184(43):V02220134. Danish. PMID 36331169
- [Background] Andersen CW, Kristensen MT. Performance Stability and Interrater Reliability of Culturally Adapted 10-Meter Walking Test for Danes with Neurological Disorders. J Stroke Cerebrovasc Dis. 2019 Sep;28(9):2459-2467. doi: 10.1016/j.jstrokecerebrovasdis.2019.06.021. Epub 2019 Jul 4. PMID 31281111
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Kristensen MT, Bandholm T, Foss NB, Ekdahl C, Kehlet H. High inter-tester reliability of the new mobility score in patients with hip fracture. J Rehabil Med. 2008 Jul;40(7):589-91. doi: 10.2340/16501977-0217. PMID 18758678
- [Background] Kristensen MT, Kehlet H. Most patients regain prefracture basic mobility after hip fracture surgery in a fast-track programme. Dan Med J. 2012 Jun;59(6):A4447. PMID 22677245
- [Background] Kempen GI, Yardley L, van Haastregt JC, Zijlstra GA, Beyer N, Hauer K, Todd C. The Short FES-I: a shortened version of the falls efficacy scale-international to assess fear of falling. Age Ageing. 2008 Jan;37(1):45-50. doi: 10.1093/ageing/afm157. Epub 2007 Nov 20. PMID 18032400
- [Background] Sorensen J, Davidsen M, Gudex C, Pedersen KM, Bronnum-Hansen H. Danish EQ-5D population norms. Scand J Public Health. 2009 Jul;37(5):467-74. doi: 10.1177/1403494809105286. Epub 2009 Jun 17. PMID 19535407
- [Background] Wittrup-Jensen KU, Lauridsen J, Gudex C, Pedersen KM. Generation of a Danish TTO value set for EQ-5D health states. Scand J Public Health. 2009 Jul;37(5):459-66. doi: 10.1177/1403494809105287. Epub 2009 May 1. PMID 19411320